CLINICAL TRIAL: NCT01106612
Title: A Randomized Controlled Trial Comparing Coronary CT Angiography and Radionuclide Stress Myocardial Perfusion Imaging in Symptomatic Inpatients With Known Coronary Artery Disease
Brief Title: Study Comparing CT Scan and Stress Test in Patients With Known Coronary Artery Disease Hospitalized for Chest Pain
Acronym: PROSPECT-CAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Jeffrey Levsky, Associate Director of Research, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMC-07-07-197-a26
Record Dates: First submitted 2010-04-12; First posted 2010-04-20 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Unstable Angina; Acute Coronary Syndrome
Keywords: randomized controlled trial; controlled clinical trial; comparative effectiveness research; chest pain; angina pectoris; non-invasive cardiac imaging; nuclear stress testing; coronary CT angiography; coronary catheterization; coronary revascularization
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial coronary CT angiography (Experimental): EKG-gated, computed tomography angiography of the coronary arteries during heart rate control
  Interventions: Procedure: Coronary CT angiography
- Initial nuclear stress test (Active Comparator): Stress radionuclide myocardial perfusion imaging
  Interventions: Procedure: Myocardial perfusion imaging

INTERVENTIONS:
Procedure: Coronary CT angiography — EKG-gated, computed tomography angiography of the coronary arteries during heart rate control
  Other Names: Coronary CTA; Coronary CT; CTA of the coronary arteries; CT of the coronary arteries; CTA; CCTA; Cardiac CTA; Cardiac CT; CT Angiography of the coronary arteries; Computed tomography angiography of the coronary arteries
  Arms: Initial coronary CT angiography
Procedure: Myocardial perfusion imaging — Stress radionuclide myocardial perfusion imaging
  Other Names: MPI; MPS; stress MPI; stress MPS; radionuclide MPI; stress nuclear; nuclear stress; nuclear stress test; nuclear stress testing; nuclear cardiology; nuclear perfusion imaging; nuclear myocardial perfusion imaging; myocardial perfusion
  Arms: Initial nuclear stress test

SUMMARY:
The purpose of this study is to determine whether coronary artery CT scanning or nuclear stress testing is better at diagnosing chest pain patients with known coronary artery disease to select appropriate candidates for coronary catheterization and re-vascularization.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted for chest pain / pressure or other suggestive symptoms
* patient has known coronary artery disease (with or without prior revascularization)
* patient has clinical need for non-invasive cardiac evaluation

Exclusion Criteria:

* evidence of ongoing myocardial infarction or hemodynamic instability
* ischemia on EKG (greater than 1mm ST segment deviation)
* contraindications to CT scanning with iodinated intravenous contrast (including allergies, asthma and renal dysfunction)
* heart rhythm precluding EKG gating
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants that undergo subsequent cardiac catheterization but do not have consequent coronary angioplasty, stenting or bypass | 3 months

SECONDARY OUTCOMES:
Length of hospital stay (time to discharge) | 1 month
Number of participants that have a subsequent non-fatal myocardial infarction | 1 year
Number of participants that die due to any cause | 1 year
Number of participants that experience a procedural complication due to non-invasive imaging, cardiac catheterization or coronary revascularization | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda B Haramati, MD, MS, Study Director — Montefiore Medical Center/Albert Einstein College of Medicine; Jeffrey M Levsky, MD, PhD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States